CLINICAL TRIAL: NCT03892109
Title: Clinical Comparative Evaluation of Different Retraction Systems in Gingival Displacement and Their Influence on Periodontal Health
Brief Title: Evaluation of Different Gingival Retraction Systems on Gingival Displacement and Periodontal Health
Acronym: retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asma Serag, Lecturer of periodontology, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000019
Record Dates: First submitted 2019-03-20; First posted 2019-03-27 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Gingival Hemorrhage
MeSH Terms: conditions — Gingival Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: unkown the group during recording the results of outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gingitrac (Active Comparator): The gingitrac cartridge was attached to the automixing gun and then the mixing syringe with intraoral tip was placed into the gingival sulcus and gingival retraction material was applied all around the selected abutment. After injecting the retraction material ,the corresponding comprecap was placed on to the abutment to push the material deep into the gingival sulcus. After 4 min, the comprecap with the set retraction material attached to it was removed from the patient mouth.
  Interventions: Other: No Cord impression material; Device: cord; Other: Gingitrac
- traxodent (Active Comparator): The traxodent cartridge was attached to the automixing gun and then the mixing syringe with intraoral tip was placed into the gingival sulcus and gingival retraction material was applied all around the tooth. After injecting the retraction material ,the corresponding comprecap was placed on to the abutment to push the material deep into the gingival sulcus. After 4 min, the comprecap with the set retraction material attached to it was removed from the patient mouth.
  Interventions: Other: No Cord impression material; Device: cord; Other: Gingitrac
- Ultrapk cord (Experimental): the cord packed into the gingival sulcus around the tooth
  Interventions: Other: No Cord impression material; Device: cord; Other: Gingitrac
- nocord (Placebo Comparator): used directly in the tray
  Interventions: Other: No Cord impression material; Device: cord; Other: Gingitrac

INTERVENTIONS:
Other: No Cord impression material — the no cord self- retracting impression material placed directly in the tray
Device: cord — Cords were placed in the gingival sulcus with use of a cord packer, and left in situ for 10 min before making the impression. None of the retraction cords were immersed in any solution or medicaments prior to insertion.
Other: Gingitrac — packed into the sulcus

SUMMARY:
The interrelationship of restorative dentistry and periodontics is a dynamic one. The interactions between restorative dentistry and periodontal health have been well-documented both clinically and histologically.

The interplay between periodontics and restorative dentistry is present at many fronts, including location of restorative margins, alloy sensitivity, crown contours, and response of the gingival tissues to restorative preparations.

Periodontal tissues form the foundation for proper esthetics, function, and comfort of the dentition, as well as the periodontal health at the restorative gingival interface consider as prerequisite for successful outcome.

Success of fixed prosthodontics restorations is largely dependent upon the long term health and stability of the surrounding periodontal structures.

The purpose of the present study was to evaluate the clinical efficacy of 4 new gingival retraction systems; traxodent, Gingitrac, Nocord, and cord , on the basis of the time taken for placement, hemorrhage control ,the amount of horizontal gingival displacement and periodontal parameter (PI, GI, CAL and PD).

DETAILED DESCRIPTION:
The interplay between periodontics and restorative dentistry is present at many fronts, including location of restorative margins, alloy sensitivity, crown contours, and response of the gingival tissues to restorative preparations.

And from fixed prothodontic point of view there are several factors affect the success and durability of restorations. In general, the type of impression making, setting accuracy, material flow, temperature, humidity, mixing, disinfection and pouring time have effects on the final accuracy of the indirect restorations. Supra-gingival margins are effective in periodontal health maintenance, but do not provide optimal aesthetics.

The primary factor in defective record of marginal details is due to the inefficacy of the gingival displacement technique.

Traditionally, procedures for soft-tissue management and isolation are classified into three main approaches: Mechanical, chemical or surgical.

material and method:-

40 subjects were selected requiring fixed prosthesis according to inclusion and exclusion criteria.

The 4 gingival retraction systems were used on the prepared abutments randomly. The time taken for placement of each retraction system was recorded.

Hemorrhage score will be recoreded. The horizontal retraction was measured on polyether impressions made before the retraction and after retraction using stereoscope.

The periodontal parameter (PI, GI, CAL and PD) will be recorded pre-operative, 1 day post-operative and 7 days post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. forty patients whose ages more than 18 years were selected requiring fixed prosthesis with minimum of two abutments.
2. Clinically and radiographically healthy gingiva and periodontium around the abutments.
3. Abutment teeth of normal size and contour (no developmental anomaly or regressive age changes).

Exclusion Criteria:

1. Age <18 years.
2. Gingival and periodontal disease.
3. Uncontrolled diabetes, hypertension, hyperthyroidism and other cardiovascular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Time of placement | the time recorded in seconds (from 1 second to 2 minutes)
  time taken for placement of each retraction system was recorded during application
Hemorrhage score | from base line to 1 day
  the amount of bleedingbleeding on probing scoring as 0, 1, and 2 (0 - no bleeding, 1 - bleeding controlled within 1 minute, bleeding, 2 - bleeding not controlled within 1 minute)

SECONDARY OUTCOMES:
Horizontal gingival displacement | from baseline to 24 hours
  The horizontal displacement was measured on polyether impressions made before the retraction and after retraction using steroscope.
Gingival index | at baseline ,after 1 day and after seven days
  according to gingival index, scored as 0,1,2 and 3( 0 = no inflamation and no gingival bleeding, 1= mild redness of the gingiva, no bleeding, 2=moderate inflammation and redness of the gingiva, edema and bleeding,3= marked redness, edema, ulceration and severe bleeding).
Pocket depth | at baseline, after 1 day and after seven days
  according to pocket depth The probe was held with a light grasp and pointed towards the apex buccally while being parallel to the long axis of the tooth. Each measurement was rounded to the lowest whole millimetre.
  according to pocket depth The probe was held with a light grasp and pointed towards the apex buccally while being parallel to the long axis of the tooth. Each measurement was rounded to the lowest whole millimetre.
Plaque index | at baseline, after 1 day and after seven days
  according to the plaque index, plaque index scoring as 0, 1, 2, and 3 (0 - no plaque and 1 - a film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or using the probe on the tooth surface, 2 - moderate accumulation of soft deposits within the gingival pocket or the tooth and gingival margin which can be seen with the naked eye, and 3 - abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided